CLINICAL TRIAL: NCT05621083
Title: Effects of Omega-3 Fatty Acids on Fasting and Postprandial TG Response in Healthy Subjects (Omega-3PT) - a Pilot Study
Brief Title: Omega-3 Fatty Acids on Fasting and Postprandial Triglycerides (TG) Response - a Pilot Study
Acronym: Omega 3-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Throne-Holst Foundation for Nutrition Research (Unknown); Horizon 2020 - European Commission (Other); GC Rieber VivoMega AS (Unknown)
Responsible Party: Principal Investigator, Stine Marie Ulven, Head of Department of Nutrition, Principal Investigator, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: REK sør-øst B 482316
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Postprandial TG response
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Start with control oil (HOSO) or start with fish oil, and then change after 12 weeks of wash out.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The principal investigator will have access to the randomization code containing the order of the oils (starting with HOSO or starting with fish oil), which is generated by an external statistician. The PI will make sure that the identical boxes with capsules (both HOSO and fish oil) will be marked only with Identification (ID) number and period number (cross over 1 and 2). The participant, the care provider and the outcomes assessor will not know the randomization code before after the data of the primary outcome has been analyzed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil (the omega-3 fatty acid supplement) (Experimental): Participants will be randomized to either start to receive fish oil (the omega-3 fatty acid supplement) for 6 weeks. Followed by a wash-out period of a minimum of 12 weeks before the treatment is changed.
  Once the classical Randomized Controlled Trial (RCT) has finished, all the participants will repeat the fish oil intervention period (adaptive design) to determine if those the investigators defined as responders continue to be defined in the same category.
  Interventions: Dietary Supplement: Omega- 3
- High-oleic sunflower oil (HOSO) containing no omega-3 fatty acids (Placebo Comparator): Participants will be randomized to either start to receive high-oleic sunflower oil (HOSO) for 6 weeks. Followed by a wash-out period of minimum 12 weeks, before the treatment is changed.
  Interventions: Dietary Supplement: HOSO

INTERVENTIONS:
Dietary Supplement: Omega- 3 — In the fish oil supplement period, the participants will receive concentrated fish oil which is equal to in total 2.3 g EPA+DHA per day during 6 weeks.
  Arms: Fish oil (the omega-3 fatty acid supplement)
Dietary Supplement: HOSO — In the HOSO period, the participants will receive similar amount of HOSO per day during 6 weeks.
  Arms: High-oleic sunflower oil (HOSO) containing no omega-3 fatty acids

SUMMARY:
The aim of this project is to elucidate how repeated exposure with omega-3 fatty acid supplementation for 6 weeks affect mean and individual fasting lipids and inflammatory responses and postprandial TG after a high fat meal with butter (50 g fat) in healthy subjects.

DETAILED DESCRIPTION:
The investigators aim to perform a randomized controlled crossover trial where each participant will act as his or her own control. Participants will be randomized to either start to receive fish oil (the omega-3 fatty acid supplement, dose of 2.3 g Eicosapentaenoic acid fatty acids (EPA) + Docosahexaenoic acid fatty acids (DHA) /day) for 6 weeks or a high-oleic sunflower oil (HOSO) containing no omega-3 fatty acids, as control followed by a wash-out period of minimum 12 weeks, before the treatment is changed for 6 weeks. Before and after each intervention period we will take fasting blood samples and collect spot morning urine. At home, the participant will perform a voluntary postprandial meal test with 61 g butter (containing 50 g fat), use DBS to collect fasting (0 h) 2, 4, 6, and 8 h blood samples after intake of the meal to measure TG which has been validated previously.

The investigators will use first part of the trial to define fasting and postprandial TG responders and non-responders. The investigators will also monitor at home the postprandial TG response to HOSO to see the participants' postprandial response to a control oil without omega-3 fatty acids. After a 12 week wash-out period, we will then repeat the fish oil intervention period once more for all in order to see if those we defined as responders continue to be defined in the same category in the repeated fish oil intervention (adaptive design). The investigators will collect exposure data, including dietary intake, physical activity, and clinical data such as BMI, body composition (such as fat mass, visceral fat, fat free mass), blood pressure, lipids and glucose and specific single nucleotide polymorphism (SNPs) to understand the impact of these factors on the individual postprandial TG response. In addition, the investigators will collect feces samples before taken before each meal test day for gut microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5-30 kg/m2
* Fasting TG level at ≥0.9 mmol/L
* Max eating one portion of fatty fish per week.
* All subjects must be willing to take two capsules with either fish oil or HOSO.
* They all need to accept to avoid taking omega-3 supplementation.
* If they use omega-3 supplements, they should wait 12 weeks before starting the study.

Exclusion Criteria:

* Unable to give informed consent
* BMI <18.5 and >30 kg/m2
* Weight change of ± 5 % of body weight in the last three months
* TG <0.9 mmol/L and > 1.7 mmol/L
* C reactive protein (CRP) >10 mg/L
* Total cholesterol >6.9 mmol/L for subjects 30-49 years and >7.8 mmol/L for subjects ≥50 years old
* Blood pressure >160/100 mm Hg
* Comorbidities including diabetes type I and II (blood glucose ≥7 mmol/L fasting), Cardiovascular diseases(CVD)/Coronary heart disease (CHD), haemophilia, anaemia (hemoglobin <120 gram/L), gastro intestinal disease, hyperthyroidism (TSH >4 Milliunits per litre (mU/L)) or inflammatory diseases such as rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), polymyalgia and other connective tissue diseases.
* Pregnant or lactating
* Having CVD/CHD or cancer past 1 year
* Allergic or intolerant to gluten, milk protein and/or lactose
* Use of medications affecting lipids and lipid metabolism, blood clotting or inflammation.
* Unwilling to separate any use of omega-3 fatty acid supplements and other supplements during the study, and fish intake more than one portion per week, 12 weeks prior to and during the study period
* Hormone treatment (stabile dose of contraception or thyroxin for the last three months excepted)
* Use of medications affecting lipids and lipid metabolism, blood clotting or inflammation. Stable dose (more than 3 months) of statin, estrogen or blood pressure medications during the trial is allowed.
* Blood donation two months prior to or during the study period
* Tobacco smoking and snuff

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Fasting TG | up to 6 weeks
  Baseline levels of circulating triglycerides

SECONDARY OUTCOMES:
Postprandial TG | up to 6 weeks
  At home, the participant will perform a voluntary postprandial meal test with 61 g butter (containing 50 g fat), use DBS to collect fasting(0 h) 2, 4, 6, and 8 h blood samples after intake of the meal
Fasting cholesterol, free fatty acids (FFA), LDL cholesterol, high-density lipoprotein (HDL) cholesterol, Apo A1, Apo B, Apo B-48 and Apo C-III, and lipoprotein subclasses, glucose and insulin | up to 6 weeks
  measure fasting levels -compare fasting levels before and after intake of omega-3 or HOSO
Fasting plasma cytokines, acute phase proteins and soluble adhesion molecules | up to 6 weeks
  measure fasting levels of all inflammatory markers before and after intake of omega-3 or HOSO
Fasting whole genome Peripheral Blood Mononuclear Cells (PBMC) transcriptome (mRNA and miRNA) | up to 6 weeks
  fasting levels before and after intake of omega-3 or HOSO
Fasting epigenome in PBMCs | up to 6 weeks
  fasting levels before and after intake of omega-3 or HOSO
Fasting targeted and non-targeted metabolic profiling in plasma | up to 6 weeks
  fasting levels before and after intake of omega-3 or HOSO
Targeted and untargeted metabolomics of spot urine to measure dietary intake biomarkers | up to 6 weeks
  Measure food intake metabolites in spot urine
SNPs in whole blood | Measured once at baseline
  measure specific SNPs related to omega-3 intake and TG response
Composition of the gut microbiome (both metabolites and bacteria composition) | up to 6 weeks
  measure metabolites in blood and feces and bacteria composition in feces

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway